CLINICAL TRIAL: NCT06549192
Title: Autonomic Responses of Amateur Child Athletes to Aerobic Exercise Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Emine Nacar, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/05-47
Record Dates: First submitted 2024-08-04; First posted 2024-08-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Heart Rate Variability; Sport

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Boxers (Active Comparator): Before the assessment begins, the children will be asked whether they have consumed any beverages containing theine and caffeine, such as tea, coffee, cola and energy drinks, which can affect the heart, in the last two hours. If this is the case, the shooting will be postponed to the next day without consuming such beverages. Participants will first have their information recorded on the general evaluation form. Their resting heart rate variability, blood pressure, heart rate and respiratory function will then be measured. After these initial measurements at rest, the participants will be given a 20 meter shuttle run test. At the end of the test, the participant will be taken to the first assessment room for a second assessment. Here, ECG, blood pressure and heart rate, spirometer measurements will be repeated. All outcome measurements will be recorded on the evaluation form.
  Interventions: Other: 20 meter shuttle run test
- Group 2: Weightlifters (Active Comparator): Before the assessment begins, the children will be asked whether they have consumed any beverages containing theine and caffeine, such as tea, coffee, cola and energy drinks, which can affect the heart, in the last two hours. If this is the case, the shooting will be postponed to the next day without consuming such beverages. Participants will first have their information recorded on the general evaluation form. Their resting heart rate variability, blood pressure, heart rate and respiratory function will then be measured. After these initial measurements at rest, the participants will be given a 20 meter shuttle run test. At the end of the test, the participant will be taken to the first assessment room for a second assessment. Here, ECG, blood pressure and heart rate, spirometer measurements will be repeated. All outcome measurements will be recorded on the evaluation form.
  Interventions: Other: 20 meter shuttle run test
- Group 3: Taekwondo players (Active Comparator): Before the assessment begins, the children will be asked whether they have consumed any beverages containing theine and caffeine, such as tea, coffee, cola and energy drinks, which can affect the heart, in the last two hours. If this is the case, the shooting will be postponed to the next day without consuming such beverages. Participants will first have their information recorded on the general evaluation form. Their resting heart rate variability, blood pressure, heart rate and respiratory function will then be measured. After these initial measurements at rest, the participants will be given a 20 meter shuttle run test. At the end of the test, the participant will be taken to the first assessment room for a second assessment. Here, ECG, blood pressure and heart rate, spirometer measurements will be repeated. All outcome measurements will be recorded on the evaluation form.
  Interventions: Other: 20 meter shuttle run test
- Group 4: Swimmer (Active Comparator): Before the assessment begins, the children will be asked whether they have consumed any beverages containing theine and caffeine, such as tea, coffee, cola and energy drinks, which can affect the heart, in the last two hours. If this is the case, the shooting will be postponed to the next day without consuming such beverages. Participants will first have their information recorded on the general evaluation form. Their resting heart rate variability, blood pressure, heart rate and respiratory function will then be measured. After these initial measurements at rest, the participants will be given a 20 meter shuttle run test. At the end of the test, the participant will be taken to the first assessment room for a second assessment. Here, ECG, blood pressure and heart rate, spirometer measurements will be repeated. All outcome measurements will be recorded on the evaluation form.
  Interventions: Other: 20 meter shuttle run test

INTERVENTIONS:
Other: 20 meter shuttle run test — 20 Meter Shuttle Run Test: Subjects run distance of 20 meters round trip. Running speed is monitored at certain intervals with help of a tape recorder that gives a signal. Subjects start running when they hear first beep and must reach other line(one foot must cross the line) by second beep. When they hear second signal, they return to starting line. The speed, which is slow at beginning, gradually increases every 10 seconds. The subject adjusts his/her pace so that he/she is on the other line at the second signal. If subject misses one signal and catches second signal, test continues. If subject misses two signals in row and doesn't reach line at other signal, test is terminated. At end of test, aerobic power values are calculated from VO2max estimation table in ml/kg/min according to number of sit-ups run. At end of test, marks obtained by athlete are calculated and VO2max value of subject is calculated in ml/kg/min from evaluation table.

SUMMARY:
The aim of our study was to investigate the relationship between aerobic capacity, which will be revealed by aerobic exercise test, and HRV, blood pressure, heart rate and pulmonary function parameters in healthy children interested in different sports branches (boxing, weightlifting, taekwando, swimming). The main questions it aims to answer are:

* Is there any relationship between aerobic capacity demonstrated by 20 m shuttle test and heart rate variability, blood pressure, heart rate and respiratory parameters in different sports branches?
* Is there a relationship between the month/year that children/adolescents are involved in sports and HRV, blood pressure and respiratory parameters?

Participants:

* Before the exercise test, ECG, blood pressure, heart rate and pulmonary function test will be performed.
* A 20 meter shuttle run test will be performed.
* Measurements will be repeated after the exercise test.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years old, registered to a club in boxing, weightlifting, taekwando and swimming (4 groups), children and adolescents who have been actively participating in their training for at least 3 months

Exclusion Criteria:

* People with neurological, orthopedic, cardiovascular diseases, those with any acute or chronic illness, smokers or drug users, elite level athletes

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
FVC | 1 hours
  A portable spirometer device will be used for the measurement of pulmonary function. During the test, the child will be placed in an upright sitting position with the pelvis in the most neutral position. Before the test, the child will be trained, demonstrated and explained what to do during the test. A different mouthpiece will be used for each child. The nose will be closed with the help of a clothespin and the measurement will be repeated 3 times and the best result will be taken into consideration. During the test, first inhale and exhale into the spirometer mouthpiece at normal tidal volume. Then a deep breath is taken and a rapid deep exhalation is requested. The exhalation period should last at least 6 s without interruption.
FEV1 | 1 hours
  A portable spirometer device will be used for the measurement of pulmonary function. During the test, the child will be placed in an upright sitting position with the pelvis in the most neutral position. Before the test, the child will be trained, demonstrated and explained what to do during the test. A different mouthpiece will be used for each child. The nose will be closed with the help of a clothespin and the measurement will be repeated 3 times and the best result will be taken into consideration. During the test, first inhale and exhale into the spirometer mouthpiece at normal tidal volume. Then a deep breath is taken and a rapid deep exhalation is requested. The exhalation period should last at least 6 s without interruption.
FEV1/FVC | 1 hours
  A portable spirometer device will be used for the measurement of pulmonary function. During the test, the child will be placed in an upright sitting position with the pelvis in the most neutral position. Before the test, the child will be trained, demonstrated and explained what to do during the test. A different mouthpiece will be used for each child. The nose will be closed with the help of a clothespin and the measurement will be repeated 3 times and the best result will be taken into consideration. During the test, first inhale and exhale into the spirometer mouthpiece at normal tidal volume. Then a deep breath is taken and a rapid deep exhalation is requested. The exhalation period should last at least 6 s without interruption.
FEF25 | 1 hours
  A portable spirometer device will be used for the measurement of pulmonary function. During the test, the child will be placed in an upright sitting position with the pelvis in the most neutral position. Before the test, the child will be trained, demonstrated and explained what to do during the test. A different mouthpiece will be used for each child. The nose will be closed with the help of a clothespin and the measurement will be repeated 3 times and the best result will be taken into consideration. During the test, first inhale and exhale into the spirometer mouthpiece at normal tidal volume. Then a deep breath is taken and a rapid deep exhalation is requested. The exhalation period should last at least 6 s without interruption.
FEF75 | 1 hours
  A portable spirometer device will be used for the measurement of pulmonary function. During the test, the child will be placed in an upright sitting position with the pelvis in the most neutral position. Before the test, the child will be trained, demonstrated and explained what to do during the test. A different mouthpiece will be used for each child. The nose will be closed with the help of a clothespin and the measurement will be repeated 3 times and the best result will be taken into consideration. During the test, first inhale and exhale into the spirometer mouthpiece at normal tidal volume. Then a deep breath is taken and a rapid deep exhalation is requested. The exhalation period should last at least 6 s without interruption.
FEF2575 | 1 hours
  A portable spirometer device will be used for the measurement of pulmonary function. During the test, the child will be placed in an upright sitting position with the pelvis in the most neutral position. Before the test, the child will be trained, demonstrated and explained what to do during the test. A different mouthpiece will be used for each child. The nose will be closed with the help of a clothespin and the measurement will be repeated 3 times and the best result will be taken into consideration. During the test, first inhale and exhale into the spirometer mouthpiece at normal tidal volume. Then a deep breath is taken and a rapid deep exhalation is requested. The exhalation period should last at least 6 s without interruption.
PEF | 1 hours
  A portable spirometer device will be used for the measurement of pulmonary function. During the test, the child will be placed in an upright sitting position with the pelvis in the most neutral position. Before the test, the child will be trained, demonstrated and explained what to do during the test. A different mouthpiece will be used for each child. The nose will be closed with the help of a clothespin and the measurement will be repeated 3 times and the best result will be taken into consideration. During the test, first inhale and exhale into the spirometer mouthpiece at normal tidal volume. Then a deep breath is taken and a rapid deep exhalation is requested. The exhalation period should last at least 6 s without interruption.
SDNN (msn) | 1 hours
  HRV obtained by electrocardiography (ECG) recording is a method that provides information about sympatho-vagal balance, calculated on the basis of the variability of the intervals between heart beats. Recordings will be taken in a quiet and calm room in the supine position. A 3-way bipolar limb lead with remote bluetooth connection (poly-spectrum-8/ex) will be used for ECG recording. Electrodes will be appropriately attached to the wrists and ankles. Participants will be asked to remove any metal objects (coins, belts, watches, bracelets, phones, etc.) that may interfere with the ECG. Participants will be pre-informed not to move, talk, breathe normally and remain in a supine position during the recording. After 5 minutes of ECG recordings are taken, data on HRV parameters will be obtained with device-specific software.
RMSSD (msn) | 1 hours
  HRV obtained by electrocardiography (ECG) recording is a method that provides information about sympatho-vagal balance, calculated on the basis of the variability of the intervals between heart beats. Recordings will be taken in a quiet and calm room in the supine position. A 3-way bipolar limb lead with remote bluetooth connection (poly-spectrum-8/ex) will be used for ECG recording. Electrodes will be appropriately attached to the wrists and ankles. Participants will be asked to remove any metal objects (coins, belts, watches, bracelets, phones, etc.) that may interfere with the ECG. Participants will be pre-informed not to move, talk, breathe normally and remain in a supine position during the recording. After 5 minutes of ECG recordings are taken, data on HRV parameters will be obtained with device-specific software.
pNN50 (%) | 1 hours
  HRV obtained by electrocardiography (ECG) recording is a method that provides information about sympatho-vagal balance, calculated on the basis of the variability of the intervals between heart beats. Recordings will be taken in a quiet and calm room in the supine position. A 3-way bipolar limb lead with remote bluetooth connection (poly-spectrum-8/ex) will be used for ECG recording. Electrodes will be appropriately attached to the wrists and ankles. Participants will be asked to remove any metal objects (coins, belts, watches, bracelets, phones, etc.) that may interfere with the ECG. Participants will be pre-informed not to move, talk, breathe normally and remain in a supine position during the recording. After 5 minutes of ECG recordings are taken, data on HRV parameters will be obtained with device-specific software.
TP (msn²) | 1 hours
  HRV obtained by electrocardiography (ECG) recording is a method that provides information about sympatho-vagal balance, calculated on the basis of the variability of the intervals between heart beats. Recordings will be taken in a quiet and calm room in the supine position. A 3-way bipolar limb lead with remote bluetooth connection (poly-spectrum-8/ex) will be used for ECG recording. Electrodes will be appropriately attached to the wrists and ankles. Participants will be asked to remove any metal objects (coins, belts, watches, bracelets, phones, etc.) that may interfere with the ECG. Participants will be pre-informed not to move, talk, breathe normally and remain in a supine position during the recording. After 5 minutes of ECG recordings are taken, data on HRV parameters will be obtained with device-specific software.
LF (msn²), %LF, LFnorm | 1 hours
  HRV obtained by electrocardiography (ECG) recording is a method that provides information about sympatho-vagal balance, calculated on the basis of the variability of the intervals between heart beats. Recordings will be taken in a quiet and calm room in the supine position. A 3-way bipolar limb lead with remote bluetooth connection (poly-spectrum-8/ex) will be used for ECG recording. Electrodes will be appropriately attached to the wrists and ankles. Participants will be asked to remove any metal objects (coins, belts, watches, bracelets, phones, etc.) that may interfere with the ECG. Participants will be pre-informed not to move, talk, breathe normally and remain in a supine position during the recording. After 5 minutes of ECG recordings are taken, data on HRV parameters will be obtained with device-specific software.
HF (msn²), %HF, HFnorm | 1 hours
  HRV obtained by electrocardiography (ECG) recording is a method that provides information about sympatho-vagal balance, calculated on the basis of the variability of the intervals between heart beats. Recordings will be taken in a quiet and calm room in the supine position. A 3-way bipolar limb lead with remote bluetooth connection (poly-spectrum-8/ex) will be used for ECG recording. Electrodes will be appropriately attached to the wrists and ankles. Participants will be asked to remove any metal objects (coins, belts, watches, bracelets, phones, etc.) that may interfere with the ECG. Participants will be pre-informed not to move, talk, breathe normally and remain in a supine position during the recording. After 5 minutes of ECG recordings are taken, data on HRV parameters will be obtained with device-specific software.
LF/HF (msn²) | 1 hours
  HRV obtained by electrocardiography (ECG) recording is a method that provides information about sympatho-vagal balance, calculated on the basis of the variability of the intervals between heart beats. Recordings will be taken in a quiet and calm room in the supine position. A 3-way bipolar limb lead with remote bluetooth connection (poly-spectrum-8/ex) will be used for ECG recording. Electrodes will be appropriately attached to the wrists and ankles. Participants will be asked to remove any metal objects (coins, belts, watches, bracelets, phones, etc.) that may interfere with the ECG. Participants will be pre-informed not to move, talk, breathe normally and remain in a supine position during the recording. After 5 minutes of ECG recordings are taken, data on HRV parameters will be obtained with device-specific software.
Systolic blood pressure | 1 hours
  Care will be taken to ensure that the person being measured is not cold, not in pain, not anxious, and not urinating or having a large bowel movement before the measurement. After the brachial artery is felt by hand, the cuff will be placed 2-3 cm above the antecubital fossa so that it is not too loose or tight. Care will be taken to ensure that the skin is not pinched, the palms are open and facing upwards. They will be warned not to make a fist. The cuff will be placed in the middle of the arm at the level of the heart so that the arm and heart are in the same horizontal plane. Blood pressure measurement is started with an automatic measuring device (F.Bosch, Germany). The device inflates the cuff enough to stop arterial blood flow. As the cuff deflates, it measures oscillations in the blood flow and then calculates the blood pressure using device-specific algorithms. The device also provides the heart rate in beats per minute.
Diastolic blood pressure | 1 hours
  Care will be taken to ensure that the person being measured is not cold, not in pain, not anxious, and not urinating or having a large bowel movement before the measurement. After the brachial artery is felt by hand, the cuff will be placed 2-3 cm above the antecubital fossa so that it is not too loose or tight. Care will be taken to ensure that the skin is not pinched, the palms are open and facing upwards. They will be warned not to make a fist. The cuff will be placed in the middle of the arm at the level of the heart so that the arm and heart are in the same horizontal plane. Blood pressure measurement is started with an automatic measuring device (F.Bosch, Germany). The device inflates the cuff enough to stop arterial blood flow. As the cuff deflates, it measures oscillations in the blood flow and then calculates the blood pressure using device-specific algorithms. The device also provides the heart rate in beats per minute.
Heart rate per minute | 1 hours
  Care will be taken to ensure that the person being measured is not cold, not in pain, not anxious, and not urinating or having a large bowel movement before the measurement. After the brachial artery is felt by hand, the cuff will be placed 2-3 cm above the antecubital fossa so that it is not too loose or tight. Care will be taken to ensure that the skin is not pinched, the palms are open and facing upwards. They will be warned not to make a fist. The cuff will be placed in the middle of the arm at the level of the heart so that the arm and heart are in the same horizontal plane. Blood pressure measurement is started with an automatic measuring device (F.Bosch, Germany). The device inflates the cuff enough to stop arterial blood flow. As the cuff deflates, it measures oscillations in the blood flow and then calculates the blood pressure using device-specific algorithms. The device also provides the heart rate in beats per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)